CLINICAL TRIAL: NCT01825655
Title: Effect of Long Acting Antihistamine on Opioid- Induced Pruritus: A Double-blind Placebo Controlled Study
Brief Title: Study of Using Long Acting Antihistamine to Treat Opioid Induced Itching
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Unable to recruit patients
Sponsor: Virginia Commonwealth University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HM20003779; IIS2012-003 (Other: Virginia Commonwealth University)
Record Dates: First submitted 2013-03-28; First posted 2013-04-05 (Estimated); Results first posted 2018-09-11 (Actual); Last update posted 2018-10-10 (Actual); Status verified 2018-09

CONDITIONS: Pruritus
MeSH Terms: conditions — Pruritus | interventions — Cetirizine; Sugars

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cetirizine (Active Comparator): zyrtec 10mg, oral, one time
  Interventions: Drug: Cetirizine
- Sugar pill (Placebo Comparator): Placebo, one pill, one time
  Interventions: Drug: Placebo or sugar pill

INTERVENTIONS:
Drug: Cetirizine
  Arms: Cetirizine
Drug: Placebo or sugar pill
  Arms: Sugar pill

SUMMARY:
The purpose of this study is determine if long acting antihistamine like cetirizine can help with itching induced by opioid pain medications.

ELIGIBILITY:
Inclusion Criteria:

* Children age 6-18yrs on opioids who develop pruritus and are willing to participate in the study

Exclusion Criteria:

* Children with history of chronic urticaria
* Children with other chronic pruritic condition like eczema, contact dermatitis, psoriasis
* Children with known hypersensitivity to cetirizine/zyrtec
* Children on H1 antihistamine like diphenhydramine, hydroxyzine, cetirizine, loratadine, fexofenadine, chlorpheniramine within the last 7days prior to randomization
* Children who have received Ondansetron within 24hrs prior to randomization
* Children who are on Tricyclic antidepressants
* Children who are unwilling or unable to swallow the capsule.
* Children with chronic liver or kidney disease

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 3 (Actual)
Dates: Start 2014-09; Primary Completion 2017-11 (Actual); Study Completion 2017-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Santhosh Kumar, M.D., Principal Investigator — Virginia Commonwealth University
Locations (1):
- Children's Hospital of Richmond at VCU, Richmond, Virginia, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: One other patient consented but did not qualify to begin the study.
Groups:
- Cetirizine: zyrtec 10mg, oral, one time
  Cetirizine
- Sugar Pill: Placebo, one pill, one time
  Placebo or sugar pill
Period: Overall Study
Arm/Group | Cetirizine | Sugar Pill
Started | 0 | 2
Completed | 0 | 2
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: No participants were randomized to the cetirizine group.
Groups:
- Total: Total of all reporting groups
Arm/Group | Cetirizine | Sugar Pill | Total
Number analyzed (Participants) | 0 | 2 | 2
Age, Customized [Count of Participants; unit: Participants]
  Between 6 and 21 years | 0 | 2 | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 2 | 2
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 0 | 1 | 1
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States |  | 2 | 2

OUTCOME MEASURES:

1. Primary Outcome: Change in Itch Score
Description: Itch score will be used to analyze our primary outcome. The subjects will have an itch score at baseline and compared to itch score at 3hrs post intervention. Itch score is measured on a scale of 1 to 4, with lower scores indicating less itchiness.
Time Frame: Baseline to 3 hours
Population: No participants were randomized into the cetirizine arm
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Cetirizine | Sugar Pill
Number analyzed (Participants) | 0 | 2
units on a scale |  | 1.5 [1 to 2]

ADVERSE EVENTS:
Time Frame: 12 hours
Description: No participants randomized to Cetirizine arm
Arm/Group | Cetirizine | Sugar Pill
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/2
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/2
Other Adverse Events (participants affected / at risk) | 0/0 | 0/2

LIMITATIONS AND CAVEATS:
The study had to prematurely end due to difficulty in recruiting subjects. The sample size is not large enough to do any statistical analysis.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-08-26): https://cdn.clinicaltrials.gov/large-docs/55/NCT01825655/Prot_SAP_000.pdf